CLINICAL TRIAL: NCT02991560
Title: Effects of Various Taping Techniques in Lateral Epicondylitis Administered in Addition to an Intensive Physiotherapy Program on Functional and Ultrasonographic Outcomes: a Double-blind, Randomized Controlled Study
Brief Title: Effects of Various Taping Techniques in Lateral Epicondylitis on Functional and Ultrasonographic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, GulOznur KARABICAK, Phd PT, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEK 10/83
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Tennis Elbow
Keywords: physiotherapy; taping; conservative treatment
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinesio tape (KT) (Experimental): The KT group was taped 2 days a week for 4 weeks using the muscle and fascia correction techniques
  Interventions: Other: Strengthening exercises; Other: Intensive Physioytherapy; Device: Kinesio taping
- Athletic taping (AT) (Experimental): An athletic tape with adhesive backing was used (38 mm wide-Muller Protape-The Netherlands).
  Interventions: Other: Strengthening exercises; Other: Intensive Physioytherapy; Device: Athletic taping

INTERVENTIONS:
Other: Strengthening exercises — The exercises consisted of 3 sets with 20 repetitions of wrist and elbow flexion; 2 sets with 10 repetitions of wrist extension strengthening starting with 50% of the maximum strength and density increasing the resistance each week; and finally, 2 sets with 10 repetitions of the wrist flexor and extensor muscle groups comprising 20 sec of stretching and 10 sec of relaxing using the healthy hand.
Other: Intensive Physioytherapy — The treatment consisted of a cold pack (enclosed in a moist towel for 12 minutes around the elbow joint), TENS (in an asymmetrical biphasic wave form and burst modulation, current width 150 mms, pulse frequency 5 Hz), and deep transverse friction massage (2 minutes of application to the locally sensitive areas determined through palpation on anterolateral surface of lateral epicondyle) followed by home exercises.
Device: Kinesio taping — Kinesio tape has been implemented on forearm of the patients for the treatment of lateral epicondylitis
  Other Names: KT
  Arms: Kinesio tape (KT)
Device: Athletic taping — By athletic taping, similar effects with Kinesio taping were aimed to gain. Considering the McConnel principles
  Other Names: AT
  Arms: Athletic taping (AT)

SUMMARY:
To compare the early effects of the application of elastic (Kinesio Tape®) and non-elastic (Athletic Tape) taping as part of the conventional physiotherapy of the lateral epicondylitis using the results from ultrasonography and clinical tests.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE), also known as tennis elbow, is an overuse injury causing elbow pain, and it is difficult to treat. It is characterized with frequent pain and sensitivity at the lateral section of the elbow, mostly at the extensor tendon (extensor carpi radialis brevis [ECRB]) origin and the extensor digitorum communis [EDC] muscle. It was estimated that annually it occurs in about 1%-3% of adult individuals worldwide. There is no consensus regarding its etiology; however, it has been associated with repetitive movements, smoking, and factors increasing physical load, such as obesity. In recent studies, workplace use of non-naturally positioned elbow and wrist have been associated with elbow pain. In addition, repetitive microtraumas have been known to be triggering injuries.

Pain is the primary complaint in LE patients. Pain increases with activity, and it becomes acute with injury or trauma. LE is associated with decreased extensor muscle strength and variations in biomechanics; however, it has been a matter of debate whether these variations are the cause or the result of LE. In its pathophysiology, three interacting components, namely local tendon pathology, changes in the pain system, and losses in motor function have been reported. Recent studies have highlighted that, rather than an inflammatory condition, tendinosis (chronic symptomatic degeneration of tendon) occurs in the forearm common extensor muscle tendon adhering to the lateral epicondyle of the humerus. Ultrasound evaluations indicate various tendon pathologies, such as tendon thickening, focused hypoechogenic zones, tendon lacerations, and calcification.

LE may heal on its own and usually responds to conservative treatment. In case conservative treatment is inconclusive, surgical methods may be opted for. Several conservative methods are among the treatment options for LE, such as resting, nonsteroidal anti-inflammatory drugs (NSAID), injection treatments, exercises, and physiotherapy programs involving manual therapy techniques, massage, braces, deep friction message, extracorporeal shockwave, low level laser therapy, low frequency electrical stimulation, and other electrophysiological agents. The use of non-elastic taping techniques is an approach utilized in the conservative treatment of LE and there exist reports examining its instantaneous effects on muscle strength, grip strength, and pain; however, it was indicated that further studies are warranted to show the effectiveness of taping. Kinesio Taping®, which involves elastic tapes, is rather a more recent technique used in orthopedic injuries in addition to physiotherapy, and it has been gaining popularity. Even though there are reports indicating the effects of adhesive tape on muscle and grip strength in LE patients, its effectiveness could not be compared with other treatment modalities because of several reasons, such as its instantaneous effects or the lack of a control group.

The literature review shows that, due to the structural differences between athletic tape and Kinesio Tape®, athletic taping applications are rather adopted to control the movement of the joint with pain, to support non-contractile structures, such as ligament and capsule, and for stability. Studies utilizing non-elastic tapes in the treatment of LE are inadequate because they examine effects in the acute period and they lack comparisons. On the other hand, it has been observed that Kinesio Tape® is mostly used for functional support, muscular facilitation, and myofascial relaxation, and studies focusing on the management of lateral epicondylitis are scarce.

The aim of the present study is, in LE patients, to compare the short-term effects of two different taping techniques in addition to an intense physiotherapy program on the severity of pain, grip strength, functional status, joint limitations, and structural changes in tendons that can be indicated by diagnostic USG

ELIGIBILITY:
Inclusion Criteria:

pain over the lateral epicondyle, pain during grip strength testing, pain in one of the following tests: extensor carpi radialis test

-

Exclusion Criteria:

* inflammatory, autoimmune, endocrine, or kidney diseases, cubital tunnel syndrome, carpal tunnel syndrome, radiculopathies due to cervical disc pathologies, additional shoulder-hand-wrist pathologies, inflammatory arthritis, upper extremity operations or traumas, allergies to the adhesive tape, and those who received corticosteroid injection and used any oral anti-inflammatory medicine due to lateral epicondylitis within the previous month

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
DASH | 30 days
  The patients were asked to grade the activities involving shoulder, arm, and hand motions within the previous week as "without any difficulty"

SECONDARY OUTCOMES:
Grip strength | 30 days
  Grip strength was measured using a Jamar hand dynamometer in kilograms. The measurement was performed 3 times and the mean value was used for evaluation. The patients were seated on an armless chair with 90° flexion of hip and knee. The patients grasped the dynamometer for a maximum of 3 seconds while their shoulders were in adduction-neutral rotation, their wrists were in flexion, and the forearms were in semipronation to provide a stronger grip
USG examinations | 30days
  USG examinations were performed in real-time using a GE Logiq 7 ultrasound scanner (General Electric Medical Systems, USA) with a linear 12 MHz (10-14 MHz) probe. A standard technique, as outlined by the European Society of Musculoskeletal Skeletal Radiology ultrasound subcommittee32, was employed for all tests
Muscle strength | 30days
  Muscle strength of the wrist flexion and extension was evaluated using the Biodex Multi-joint Isokinetic System 3 Pro. Measurements were performed at two different speeds: 60°/sec and 120°/sec.
Pain intensity | 30 days
  Pain intensity was evaluated using the visual analog score (VAS) at night and rest-activity. The patients assigned a value for their pain between 0 and 10 on the VAS scale. In this scale, the absence of pain was marked as 0 while the most severe unbearable pain was expressed as 10.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Bek, Proffessor, Study Director — Hacettepe University

IPD SHARING:
Plan to Share IPD: No